CLINICAL TRIAL: NCT03195582
Title: The Effect of Chlorohexidine Gel on Tissue Healing Following Surgical Exposure of Dental Implants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Hadar Zigdon MD, Dr., Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0480-16-RMB
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Implant Infection; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: patients will be divided randomly in to 2 groups:
  1. Control: following uncovering of the implant a 4 mm height healing abutment will be screwed to the implant (the standard treatment modality) without using CHX gel or any other gel.
  2. Test group: following implant exposure this group will receive CHX 1% gel (Corsodyl®) the gel will be applied on the abutment as well as on the implant internal hex and then a 4 mm healing abutment will be connected.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study will be single blinded. The examiners of the clinical measurements, ELISA samples and the radiographs will be blinded to the patient's group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): following local anesthesia buccal and lingual flaps will be raised minimally, the cover screw will be removed from the implant .In the test group, Corsodyl gel 1% Chlorohexidine will be applied on the implant and the healing abutment. Healing abutment of 4 mm height will be screwed to the implant and flap will be sutured with silk 4-0 sutures.
  Parallel radiograph will be taken after the surgery
  Interventions: Drug: Corsodyl
- CONTROL group (No Intervention): following local anesthesia buccal and lingual flaps will be raised minimally, the cover screw will be removed from the implant .In the control group, Corsodyl gel 1% Chlorohexidine will not be applied on the implant and the healing abutment). Healing abutment of 4 mm height will be screwed to the implant and flap will be sutured with silk 4-0 sutures.
  Parallel radiograph will be taken after the surgery

INTERVENTIONS:
Drug: Corsodyl — following local anesthesia buccal and lingual flaps will be raised minimally, the cover screw will be removed from the implant. In the test group, Corsodyl gel 1% CLOROHEXIDINE will be applied on the implant and the healing abutment.
  Other Names: Test group
  Arms: Test group

SUMMARY:
The aim of this study is to evaluate the healing of peri-implat tissue following surgical uncovering with the adjunctive use of Chlorohexidine (CHX) gel.

DETAILED DESCRIPTION:
Patients who received implants in our department, and scheduled for surgical uncovering of the implants will be asked to participate in this clinical trial (40) Patients from Department of periodontology, Rambam Health campus, Haifa in Israel will be recruited to Randomized clinical trial; patients will be divided randomly in to 2 groups:

1. Control: following uncovering of the implant a 4 mm height healing abutment will be screwed to the implant (the standard treatment modality) without using Chlorohexidine gel or any other gel.
2. Test group: following implant exposure this group will receive Chlorohexidine 1% gel (Corsodyl®) the gel will be applied on the abutment as well as on the implant internal hex and then a 4 mm healing abutment will be connected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are willing to participate and willing to provide an informed consent.
2. Males and females between the ages 18-80
3. In good general health.
4. Patients who received dental implants and require implant uncovering (if there is more than 1 implant, a minimum radiographic distance of 3 mm will be required between implants).

Exclusion Criteria:

1. Uncontrolled Type 1 or type 2 diabetes patients( HbA1C>7).
2. Subjects treated for at least 2 weeks with any medication known to affect soft tissue condition within one month prior to baseline examination (e.g., Phenytoin, Cyclosporine, and chronic use of Bisphosphonates).
3. Patients who underwent guided bone regeneration during implant placement.
4. Patients who used antibiotic during the study or 4 weeks prior to the baseline.
5. Active periodontitis patients.
6. Subjects with presence of active systemic infectious diseases such as: Hepatitis, HIV, history of tuberculosis.
7. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Recession depth | 3 MONTHS
  Distance from the healing abutment top to the free gingival margin will be measured by periodontal probe at the mid-buccal aspect of the healing abutment. Recession (Rec) is defined as the difference in millimeters between baseline to to 3 months .

SECONDARY OUTCOMES:
PROBING DEPTH | 3 MONTHS
  The distance between the free gingival margin to the base of the pocket will be measured by periodontal probe in millimeters.
Width of the keratinized mucosa (WKM) | 3 MONTHS
  the distance in millimeters between the free gingival margin to the mucogingival line will be measured by periodontal probe .

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, Dr., Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No